CLINICAL TRIAL: NCT05098327
Title: Role of Pioglitazone Therapy in Management of Insulin Resistance Associated With Androgen Deprivation Therapy (ADT) in Patients With Prostate Cancer
Brief Title: Pioglitazone and Insulin Resistance in ADT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no participant enrolled due to lack of interest.
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, paresh Dandona, SUNY Distinguished Professor of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005310; UL1TR001412 (NIH)
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer; Insulin Resistance; Diabetes Mellitus, Type 2; Androgen Deficiency
MeSH Terms: conditions — Prostatic Neoplasms; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prostate cancer on ADT receiving pioglitazone (Active Comparator): Subjects will receive a 12-week supply of pioglitazone 30 mg dose 1 tab daily
  Interventions: Drug: Pioglitazone 30 mg
- Prostate cancer on ADT receiving placebo (Placebo Comparator): Subjects will receive a 12 week supply of placebo pills containing cellulose
  Interventions: Drug: Placebo
- Prostate cancer not on ADT (No Intervention): No intervention will be done in this group

INTERVENTIONS:
Drug: Pioglitazone 30 mg — pioglitazone 30 mg dose 1 tab daily will be given for 12 weeks
  Other Names: Actos
  Arms: Prostate cancer on ADT receiving pioglitazone
Drug: Placebo — placebo pills containing cellulose 1 pill daily will be given for 12 weeks
  Arms: Prostate cancer on ADT receiving placebo

SUMMARY:
This study is being done to establish the mechanisms underlying insulin resistance (reduced insulin action that can lead to high blood sugar and maybe diabetes) in patients undergoing androgen deprivation therapy (ADT) for prostate carcinoma as well as to investigate the role of pioglitazone therapy in reduction/ reversal of that insulin resistance

DETAILED DESCRIPTION:
This is a single-center, cross-sectional then prospective, randomized single-blinded study with 2 groups of subjects. One group will be men with prostate cancer in various stages of ADT and the other group will be men with prostate cancer not on ADT as control group.

Patients interested in participating who meet the inclusion/exclusion criteria and who agree to undergo blood draws and fat biopsy will be identified from the Genito-urinary oncology and urology clinics. These patients will be referred to the Diabetes and Endocrinology Research Center of WNY where they will undergo blood draws in fasting state.

On the screening day, participants will be asked to complete the informed consent, medical history and physical exam, and non-fasting blood draws (for CBC, CMP and HbA1c) prior to participating in the study. 30 ml of blood will be drawn at this visit.

Subjects who qualify and consent to take part in the study will be called in for the baseline study visit where they will undergo blood draws in fasting state. HOMA-IR method will be used to determine insulin resistance. Subcutaneous fat biopsies will be performed in all patients.

Within the ADT group, subjects will be assigned a number by a computerized simple random number generation program (Excel, Microsoft Inc.) and will be randomized (1:1) to receive either pioglitazone or placebo. The patient will be blinded to the treatment, however, the research team will not. Subjects will be given a 12 week supply of pioglitazone 30 mg or placebo pills containing cellulose that will take once a day in morning. Subjects who develop side effects (weight gain, pedal edema) on the 30 mg dose will be asked to reduce the dose to 15 mg.

Subjects will then return to the research center in 12 weeks for visit 2 where the fasting blood draws and subcutaneous fat biopsies will be performed again. The subjects will then be discharged from the study and follow with their physicians. Subject will receive a phone call after 1 and 4 weeks following start of treatment to collect any safety data. Patients will be instructed to call the research center anytime they have a question or side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age ≥18 years of age.
2. Body Mass Index of > 25 kg/m2
3. Biopsy-confirmed prostate adenocarcinoma currently on androgen deprivation therapy (ADT) for minimum of 3 months for the ADT group and biopsy-confirmed prostate adenocarcinoma not on ADT for control group

5. Hemoglobin > 11 g/dL, Creatinine < 1.5x ULN and liver function tests < 2x ULN 6. Participant must be able to read, write, and understand the English language and be able to provide written consent 7. Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

1. Known clinically significant severe COPD, ischemic heart disease, congestive heart failure, and/or significant cardiac arrhythmias
2. Any patient with known diabetes (A1c > 6.4%) or an anti-diabetic drug
3. Any condition contraindicating additional blood collection beyond standard of care
4. Subjects with known allergy to lidocaine (this is used to anesthetize area for fat biopsy)
5. Subjects with known allergy to pioglitazone or other thiazolidinediones
6. Subjects with pioglitazone use in last 6 months
7. Subjects with congestive Heart Failure Class 3 or 4
8. Subjects with osteoporosis, including history of fragility fracture
9. Subjects with history of bladder cancer
10. Subjects on chronic use of androgens, or opiates in the last 6 months or with panhypopituitarism, congenital HH (hypogonadotropic hypogonadism), prolactinoma, head trauma
11. Unwilling or unable to follow protocol requirements
12. Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to undergo study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 12 weeks
  Change in HOMA-IR (the main index for evaluating insulin resistance) following pioglitazone and placebo treatment.

SECONDARY OUTCOMES:
IRS-1 serine phosphorylation | 12 weeks
  Determine levels of IRS-1 serine phosphorylation in adipose tissue and MNC as a molecular marker of inflammation induced insulin resistance at baseline and after pioglitazone and placebo treatments
IRβ | 12 weeks
  Changes in expression of insulin signaling gene (IRβ) in both adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
IRS-1 | 12 weeks
  Changes in expression of insulin signaling gene (IRS-1) in both adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
AKT-2 | 12 weeks
  Changes in expression of insulin signaling gene (AKT-2) in both adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
GLUT-4 | 12 weeks
  Changes in expression of GLUT-4 in adipose tissue between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
TNF-α | 12 weeks
  Changes in expression of proinflammatory gene (TNF-α) that interfere with insulin signaling transduction in adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
IL 1β | 12 weeks
  Changes in expression of proinflammatory gene (IL 1β) that interfere with insulin signaling transduction in adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
IKK-β | 12 weeks
  Changes in expression of proinflammatory gene (IKK-β) that interfere with insulin signaling transduction in adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
SOCS-3 | 12 weeks
  Changes in expression of proinflammatory gene (SOCS-3) that interfere with insulin signaling transduction in adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
PTB-1B | 12 weeks
  Changes in expression of proinflammatory gene (PTB-1B) that interfere with insulin signaling transduction in adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
JNK-1 | 12 weeks
  Changes in expression of proinflammatory gene (JNK-1) that interfere with insulin signaling transduction in adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group
TLR-4 | 12 weeks
  Changes in expression of proinflammatory gene (TLR-4) that interfere with insulin signaling transduction in adipose tissue and MNC between the ADT and non-ADT groups at baseline and after pioglitazone and placebo treatments in ADT group

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, PhD, Principal Investigator — SUNY at Buffalo
Locations (1):
- Diabetes and Endocrinology Research Center of WNY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No